CLINICAL TRIAL: NCT05252026
Title: Indicated Prevention Transdiagnostic Intervention for Adolescents At High Risk of Emotional Problems
Acronym: PROCARE-I
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jaén (Other)
Collaborators: Universidad Miguel Hernandez de Elche (Other); University Rovira i Virgili (Other); University of Miami (Other)
Responsible Party: Principal Investigator, LuisJoaquin Garcia-Lopez, Full Professor, University of Jaén
Allocation: Randomized | Model: Factorial | Masking: Triple | Purpose: Prevention
Other Study IDs: UJA-PROCARE-I
Record Dates: First submitted 2022-02-11; First posted 2022-02-23 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Anxiety Disorders and Symptoms; Depressive Symptoms
Keywords: ADOLESCENCE; TRANSDIAGNOSTIC; indicated PREVENTION; Randomized-Controlled Trial; high-risk
MeSH Terms: conditions — Anxiety Disorders; Depression

STUDY DESIGN:
Intervention Model Description: One intervention is evaluated in parallel against a active control group
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PROCARE-I (UP-A for indicated purposes) (Experimental): To ensure cost-effectiveness, PROCARE-I intervention will be designed as a brief 8-session child-focused programme by adapting the core modules from UP-A, along with one individual session with adolescent and parents. Sessions will be delivered in reduced groups, using a typical indicated preventive intervention format focused on cost-effectiveness.
  Interventions: Behavioral: PROCARE-I (UP-A for indicated purposes)
- Active control condition (Experimental): The active control condition will be based on the "U talk programme" developed by Prf. Jill Ehrenreich-May at University of Miami and colleagues. It follows a similar structure as the UP-A original programme and allows for one alternative compare condition to PROCARE-I. The U Talk programme support-based group condition will be used as active control condition.
  Interventions: Behavioral: Active control condition

INTERVENTIONS:
Behavioral: PROCARE-I (UP-A for indicated purposes) — This intervention is meant to respond to the heterogeneity inherent in emotional difficulties presentation by extinguishing distress associated with the presentation of heightened negative emotion in general and reduction or elimination of resultant emotionally-driven behaviours, including avoidance, escape, aggression, and controlling behaviours (e.g., reassurance seeking) that reinforce emotional distress intensity over time.
  Arms: PROCARE-I (UP-A for indicated purposes)
Behavioral: Active control condition — Psychoeducation about many different emotions, emphasis on discussing thoughts, feelings, and behavior as parts of emotion, and emphasis on providing support around generally distressing events.
  Arms: Active control condition

SUMMARY:
Emotional disorders (anxiety and/or depression) are severely undiagnosed and untreated despite being among the most common mental disorders, particularly at a young age. Half of all mental disorders begin by age 14; three-quarters by age 24, which makes adolescence a particularly crucial stage. In adolescence, prodromal signs of mental disorders and even full-blown clinical conditions often remain undetected, undiagnosed and untreated. However, there is an absence of evidence-based protocols to reach at high risk youth for developing emotional disorders. There is an urgent need for a paradigm shift by developing intervention protocols to early identify and treat vulnerable adolescents, thus preventing them from developing severe mental disorders later on in life. Mental health indicated prevention is key to helping at-high risk adolescents thrive before emotional disorder evolves. To cover this gap, PROCARE-I is conceptualized as a modularized indicated preventive programme for adolescents aged 12 to 18 years, adapting UP-A protocol with author's permission and supervision. Adolescents will be allocated to a 2-arm intervention trial, delivered as a group, as telehealth format as a result of Covid19 restrictions imposed by government. The PROCARE-I protocol aims to enhance protective factors that will eventually lead to lasting positive effects for adolescents. PROCARE-I will combine quantitative analysis, with special attention to vulnerable groups in a sex/gender disaggregated way. The PROCARE-I project is expected to have a far impact ultimately contributing to preventing and reducing the prevalence of emotional disorders in the young. The outcomes of PROCARE-I will contribute to identifying and treating vulnerable adolescents at high risk for emotional mental at an early stage, before they incur personal, societal and economic cost. PROCARE-I will be culturally-adapted and implemented as a multicenter Randomized-Controlled Trial (RCT). PROCARE-I will be designed to be an acceptable, scalable, and sustainable indicated prevention program.

DETAILED DESCRIPTION:
The general objective of PROCARE-I is to design, implement and evaluate a indicated 8-session preventive group intervention for adolescents aged 12-18 at high risk of emotional disorders like anxiety and depression. The intervention will be based on the Unified protocol for transdiagnostic treatment of emotional disorders in adolescents (UP-A), already proven as effective in the US, but adapted with indicated prevention purposes in Spain thanks support of main author of the protocol (Prf. Ehrenreich-May). It will be culturally-adapted and designed to be an acceptable, scalable, and sustainable indicated prevention program. METHODOLOGY The methodology was designed in order to achieve the project's objective of treating vulnerable adolescents at high risk of developing emotional disorders. PROCARE-I working plan will be divided into 3 interconnected stages. Firstly, in order to identify adolescents at high risk of suffering emotional disorders (anxiety and depression), the following self-reports will be administered to adolescents: Strengths and Difficulties Questionnaire (SDQ) to evaluate adolescents at-risk of emotional disorders, and the Revised Child Anxiety and Depression Scale-30 (RCADS-30) will screen for presence/absence of emotional symptomatology. Finally, ADIS5-C/P will be administered to rule-out presence of anxiety and/or mood disorders. Valuing voices from stakeholders and end-users, the investigators will focus on the study of the influence of the above described variables. Third, the investigators will test a indicated preventive intervention using multi-center randomized control trial in Spain. Special attention will be paid to particularly vulnerable young people, such as disabled, refugees, immigrants, or minorities (national, ethnic, linguistic, religious, and sexual).

IMPACT The need to include mental health among the first priorities of the public health agenda has been increasingly recognized over the past decades. The outcomes of the PROCARE-I project will have a far impact ultimately contributing to preventing and reducing the prevalence of mental disorders in the young. These problems are wide-ranging, long-lasting, and enormous and impose a range of costs on individuals, families and communities. The outcomes of the project, if successful, will have far reaching implications, contributing to identifying and treating adolescents at high risk for emotional mental disorders at an early stage, before they incur personal, societal and economic cost.

ELIGIBILITY:
Inclusion Criteria:

* written informed consent from adolescent and legal guardian
* able to attend prevention modules on his/her own
* language competence
* Strengths and Difficulties Questionnaire ""probable diagnoses"
* score above cut-off for Revised Child Anxiety and Depression Scale-30
* absence of anxiety and/or mood disorders

Exclusion Criteria:

* in- or outpatient
* concomitant psychological/psychiatric treatment
* acute suicidality
* general medical contraindications that hamper attendance to prevention modules
* Strengths and Difficulties Questionnaire "unlikely" or "possible diagnoses"
* presence of mood and/or anxiety disorders

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 68 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2022-06-30 (Actual)

PRIMARY OUTCOMES:
Self-reported anxiety and mood symptomatology | Baseline to 7 months after start of interventions
  The study's primary outcome was self-reported anxiety and mood symptomatology as assessed by Revised Child Anxiety Depression Scale (RCADS-30). Total scores range from 0 to 90. Higher scores mean a worse outcome
Factors associated with adolescents' mental health | Baseline to 7 months after start of interventions
  The study's primary outcome was self-reported risk and protective factors level of emotional disorders as assessed by Strengths and Difficulties Questionnaire (SDQ). Total scores range from 0 to 50. Higher scores mean a worse outcome.
Absence of emotional disorders | Baseline to 7 months after start of interventions
  The study's primary outcome was absence of any emotional disorders over the long-term measured by the ADIS-5-C/P

SECONDARY OUTCOMES:
Health-related quality of life | Baseline to 7 months after start of interventions
  Secondary outcome assessed included self-reported changes in health-related quality of life as assessed by KIDSCREEN-10. Total scores range from 10 to 50. Higher scores mean a better outcome.
Economic evaluations | Baseline to 7 months after start of interventions
  Implementation service costs (training, program materials, provider salaries), costs to school system, and later health costs saved for preventing emotional problems that could narrow cumulative disparities in mental health and disadvantage later in life.
Psychological flexibility | Baseline to 7 months after start of interventions]
  Psychological flexibility as assessed by Willingness and Action Measure for Children and Adolescents (WAM-C/A).
  Total scores range from 0 to 56. Higher scores mean a better outcome.
Emotional regulation | Baseline to 7 months after start of interventions]
  The Difficulties in Emotion Regulation Scale (DERS)

CONTACTS AND LOCATIONS:
Overall Officials: Luis-Joaquin Garcia-Lopez, Ph.D., Principal Investigator — University of Jaen
Locations (3):
- Spain (3):
  - Universidad Miguel Hernandez, Elche, Alicante
  - University of Jaen, Jaén, Jaen
  - Universitat Rovira i Virgili, Tarragona

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Garcia-Escalera J, Valiente RM, Sandin B, Ehrenreich-May J, Prieto A, Chorot P. The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (UP-A) Adapted as a School-Based Anxiety and Depression Prevention Program: An Initial Cluster Randomized Wait-List-Controlled Trial. Behav Ther. 2020 May;51(3):461-473. doi: 10.1016/j.beth.2019.08.003. Epub 2019 Aug 14. PMID 32402261
- [Result] Sandin B, Garcia-Escalera J, Valiente RM, Espinosa V, Chorot P. Clinical Utility of an Internet-Delivered Version of the Unified Protocol for Transdiagnostic Treatment of Emotional Disorders in Adolescents (iUP-A): A Pilot Open Trial. Int J Environ Res Public Health. 2020 Nov 10;17(22):8306. doi: 10.3390/ijerph17228306. PMID 33182711
- [Result] Levin L, Henderson HA, Ehrenreich-May J. Interpersonal predictors of early therapeutic alliance in a transdiagnostic cognitive-behavioral treatment for adolescents with anxiety and depression. Psychotherapy (Chic). 2012 Jun;49(2):218-230. doi: 10.1037/a0028265. PMID 22642525
- [Result] Queen AH, Barlow DH, Ehrenreich-May J. The trajectories of adolescent anxiety and depressive symptoms over the course of a transdiagnostic treatment. J Anxiety Disord. 2014 Aug;28(6):511-21. doi: 10.1016/j.janxdis.2014.05.007. Epub 2014 Jun 2. PMID 24960439
- [Result] Bilek EL, Ehrenreich-May J. An open trial investigation of a transdiagnostic group treatment for children with anxiety and depressive symptoms. Behav Ther. 2012 Dec;43(4):887-97. doi: 10.1016/j.beth.2012.04.007. Epub 2012 May 1. PMID 23046789
- [Result] Ehrenreich-May J, Rosenfield D, Queen AH, Kennedy SM, Remmes CS, Barlow DH. An initial waitlist-controlled trial of the unified protocol for the treatment of emotional disorders in adolescents. J Anxiety Disord. 2017 Mar;46:46-55. doi: 10.1016/j.janxdis.2016.10.006. Epub 2016 Oct 17. PMID 27771133